CLINICAL TRIAL: NCT04492943
Title: To Observe Whether Isoflurane Can Treat COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Zhongcong Xie, Principle Investigator, Massachusetts General Hospital
Other Study IDs: 2020P001048
Record Dates: First submitted 2020-04-24; First posted 2020-07-30 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: COVID-19
Keywords: Mechanical ventilation; Anesthesia
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood may be collected from patients if available from excess clinical blood draws conducted during routine clinical care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a blood collection and retrospective data collection study. The investigators plan to assess whether the sedative drug, isoflurane, can treat COVID-19 patients relatively better compared to other sedative drugs given during routine treatment to patients on mechanical ventilation. The investigators will also use nanoneedle biosensors to quickly detect blood IgM/IgG ratio in those patients, and (3) to establish a pre-clinical system to determine the effects of inhalational anesthetics on amounts of SARS-CoV-2 and other viruses, and pneumoniae.

DETAILED DESCRIPTION:
There are neither effective treatments nor fast detection for COVID-19. Here the investigators propose a medical records and excess clinical material study to determine whether anesthetic isoflurane can treat COVID-19. Specifically, inhalation anesthetics, including isoflurane, inhibit the replication of an RNA virus. In addition, anesthesia machines have been used to provide mechanical ventilation for COVID-19 patients at MGH and at other hospitals. Finally, due to the shortage of intravenous anesthetic propofol, inhalation anesthetics including isoflurane, delivered by the anesthesia machine, are currently used to sedate COVID-19 patients during mechanic ventilation. Moreover, isoflurane is very economical, e.g. $6 (isoflurane) versus $1200 (propofol) per patient per day in sedating COVID-19 patients. As such, the investigators propose to use this already established system in COVID-19 patients to determine whether isoflurane, delivered to lungs, can treat COVID-19 and especially COVID-19 pneumonia. In summary, the proposed study is a low risk observation research using the already established clinical care system of COVID-19 patients and the investigators will NOT have any additional procedures required for research purpose. The investigators will also collect the left-over clinical sample and then use nanotechnology to achieve fast detection of IgM/IgG ratio as the biomarker of the progress of COVID-19 following the isoflurane or propofol sedation.

Specifically, inhalation anesthetics, including isoflurane, inhibit replication of the measles virus and other RNA virus 1,2. Severe COVID-19 patients need mechanical ventilation to support lung function. The anesthesia machine can be used to ventilate lungs in these patients in addition to regular ventilators which has already been started at MGH and other hospitals as regular ventilators are extremely limited. Clinicians have already determined the settings of these machines, including humidification, for treating COVID-19 patients and the investigators will use these predetermined settings in this study. Additionally, there is a shortage of the intravenous anesthetic propofol. As a result, inhalation anesthetics including isoflurane, delivered by the anesthesia machine, are currently used to sedate COVID-19 patients during mechanic ventilation. Moreover, isoflurane is very economical, e.g. $6 (isoflurane) versus $1200 (propofol) per patient per day in sedating COVID-19 patients. As such, the investigators propose to use this already established system in COVID-19 patients to determine whether isoflurane, delivered to lungs, can treat COVID-19 and especially COVID-19 pneumonia better than other sedatives in this retrospective data collection study. Moreover, in pre-clinical studies, the investigators propose to establish a system to determine whether inhalation anesthetics can treat virus-induced pneumonia by reducing the amount of virus, e.g., SARS-CoV-2 and influenza.

Sensitive, cost-effective and fast detection of SARS-CoV-2 is extremely critical. Currently, a real-time polymerase chain reaction (PCR) test detects the genetic material of SARS-CoV-2. However, the test has large false negatives, poses risks during specimen collection and sample handling, and takes a long time (~ 8 hours). However, in response to SARS-CoV-2, IgG is the most abundant immunoglobulin to be produced and is maintained in the body after initial exposure for a long-term response. IgM is the first immunoglobulin to be produced but is primarily detected during the early onset of disease. Therefore, SARS-CoV-2 specific IgM/IgG ratio in blood could be used as biomarker for COVID-19 prognostics (Fatma et al, medRxiv, 2020), and could also be used as a measure of drug response 3. The nanoneedle technology developed at a startup-company from Harvard University (NanoMosaic LLC) provides pg/ml-level sensitivity and 10 uL sample volume for quantification of a panel of biomarkers including SARS-CoV-2 specific IgG and IgMs in a single assay. The technology uses nanoneedle biosensors densely integrated on a silicon chip and manufactured with CMOS-compatible nanofabrication processes 4. Each nanoneedle is a label-free biosensor and changes its scattering spectrum when an antigen binds to its surface. Each analyte-specific sensing area consists of a total of ~24k nanoneedles divided into a digital region (~20k nanoneedles), an analog region (~3k nanoneedles) and a fabrication QC region (~1k nanoneedles), thus providing a wider dynamic range beyond the digital counting concentration ranges. Each single analyte area, including both digital and analog sensors, is less than 500 um. With further development, the entire assay can be finished in a half-hour on a table-top instrument with less than 10 ul blood samples, which will facilitate therapeutic development and decision making for COVID-19 and other virus-induced pneumoniae.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18 years old
* Tested positive for COVID-19
* Documented SARS-CoV-2 carriage in the nasopharyngeal sample by PCR
* Intubated for mechanical ventilation with an anesthesia machine

Exclusion Criteria:

* Patient or any their family members have any contraindication for inhalation anesthetics (e.g., malignant hyperthermia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID-19 positive patients placed on mechanical ventilation
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Survival Outcome | From the date of hospital admission until date of discharge or death of any cause, assessed up to 6 months.
  Survival outcome will be based on whether the patient either (a) recovers from COVID-19 and is discharged from the hospital or (b) does not recover from COVID-19 and passes away while in the hospital.
COVID-19 Testing Methods | From the date of hospital admission until date of discharge or death of any cause, assessed up to 6 months.
  Identifying faster COVID-19 testing methods, specifically nanoneedle biotechnology.
COVID-19 Clearance | From the date of hospital admission until date of discharge or death of any cause, assessed up to 6 months.
  COVID-19 clearance will be based on whether the patient either (a) tests negative for COVID-19 after treatment in the hospital or (b) does not test negative for COVID-19 after treatment in the hospital.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
Participant data may be shared with other researches working on similar studies. The only identifiers in data sets that will be shared are (1) hospital admission dates (MM/DD/YYYY), ICU admission dates (MM/DD/YYYY), ICU discharge dates (MM/DD/YYYY), and hospital discharge dates (MM/DD/YYYY).